CLINICAL TRIAL: NCT03912857
Title: A Study of Camrelizumab Combined With Apatinib in the Treatment of Advanced Metastatic Colorectal Cancer:One-arm, Single-center, Open-stage Phase II Clinical
Brief Title: Camrelizumab(SHR-1210) Combined With Apatinib in the Treatment of Advanced Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Ruihua Xu, Dean, Chief Physician, headof Gastroenterology, Professor，Principal Investigator, Clinical Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PD-1/mCRC
Record Dates: First submitted 2019-04-09; First posted 2019-04-11 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Metastatic Colorectal Cancer
Keywords: mCRC MSI-H
MeSH Terms: conditions — Colorectal Neoplasms | interventions — camrelizumab; apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- test group (Experimental): Drug:Camrelizumab(SHR-1210) 200mg, once every 2 weeks, each 4 weeks is 1cycle.
  Apatinib :250 mg or 375 mg, qd
  Interventions: Drug: Camrelizumab

INTERVENTIONS:
Drug: Camrelizumab — Experimental: test group Drug:Camrelizumab(SHR-1210) 200mg, once every 2 weeks, each 4 weeks is 1cycle.
  Apatinib :250 mg or 375 mg, qd
  Other Names: Apatinib

SUMMARY:
The incidence and mortality of colorectal cancer in China's cancer disease spectrum is on the rise, and it is a common malignant tumor that harms the health of Chinese residents.This study was a one-arm, single-center, open clinical study. A total of 50 patients were enrolled in the study.

DETAILED DESCRIPTION:
Because of the clinical lack of research to explore the safety and efficacy of VEGFR2 inhibitors in combination with anti-PD-1 antibodies in the treatment of colorectal cancer, we intend to conduct a single-center, one-arm, open, investigator-initiated clinical study aimed at To clarify the efficacy and tolerability of PD-1 antibody SHR-1210 in combination with VEGFR2 inhibitor apatinib in patients with metastatic colorectal cancer microsatellite stabilization, and to explore the tumor tissue and hematological immune molecular markers predicting the effectiveness of the protocol. Things. The results of this clinical trial will likely increase the objective response rate of advanced colorectal cancer after standard treatment, and hopefully find molecular markers that can predict the sensitivity of colorectal cancer PD-1 immunotherapy combined with anti-angiogenic targeted therapy. Therefore, it has important clinical significance.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily join the study and sign an informed consent form;
2. Age ≥ 18 years old and ≤ 75 years old, both men and women;
3. Colorectal cancer confirmed by histology or cytology with distant metastasis; confirmed to be a microsatellite stable patient.
4. Previously received single or combined use of oxaliplatin, irinotecan, fluorouracil, second-line and above treatment failure or inability to tolerate second-line and above treatment;
5. For neoadjuvant/adjuvant therapy (chemotherapy or chemoradiotherapy), if disease progression occurs during treatment or within 6 months of discontinuation of treatment, it should be counted as first-line treatment failure;
6. According to the solid tumor efficacy evaluation standard (RECIST1.1), at least one measurable lesion, measurable lesions should not have received local treatment such as radiotherapy (target lesions in the previous radiotherapy area, if confirmed to progress, and in line with RECIST1 .1 standard, can also be used as a target lesion.);
7. Tissue samples should be provided for molecular pathology analysis, preferably newly acquired tissues, and patients who are unable to provide newly acquired tissues can provide 10 sheets of 5um thick paraffin sections that are archived and preserved;
8. ECOG: 0 to 1 (see Annex 1);
9. Can swallow pills;
10. Expected survival ≥ 12 weeks;
11. The function of vital organs meets the following requirements (no blood components and cell growth factors are allowed for 2 weeks prior to the start of the study):Absolute neutrophil count (ANC) ≥ 1.5 × 109 / L;Platelets ≥75×109/L; Hemoglobin ≥ 8g / dL;Serum albumin ≥ 2.8g / dL;Bilirubin ≤ 1.5 times ULN, ALT and AST ≤ 2.5 times ULN; if there is liver metastasis, ALT and AST ≤ 5 times ULN; Creatinine clearance ≥ 50mL / min (Cockcroft-Gault, see Annex II);

Exclusion Criteria:

1. The subject has any active autoimmune disease or a history of autoimmune disease (such as the following, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituititis, vasculitis) , nephritis, hyperthyroidism, decreased thyroid function; subjects with vitiligo or complete remission in childhood asthma, can be included without any intervention in adults; subjects who require bronchodilators for medical intervention can not be included );
2. Subjects are using immunosuppressive agents, or systemic, or absorbable local hormonal therapies for immunosuppression purposes (dose >10 mg/day of prednisone or other therapeutic hormones) and within 2 weeks prior to enrollment Still continuing to use;
3. Severe allergic reactions to other monoclonal antibodies;
4. Subjects have clinically symptomatic central nervous system metastases (eg, cerebral edema, need for hormonal intervention, or progression of brain metastases). Previously treated with brain or meningeal metastases, such as patients with clinically stable (MRI) who have been on hold for at least 1 month and who have stopped systemic hormonal therapy (dose >10 mg/day of prednisone or other therapeutic hormones) for more than 2 weeks can be included ;
5. Suffering from high blood pressure, and can not be well controlled by antihypertensive drugs (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg);
6. There are clinical symptoms or diseases of the heart that are not well controlled, such as: (1) NYHA class 2 or higher heart failure (2) unstable angina (3) myocardial infarction within 1 year (4) clinically significant supraventricular Or ventricular arrhythmia requires treatment or intervention;
7. abnormal blood coagulation (PT>16s, APTT>43s, TT>21s, Fbg<2g/L), with bleeding tendency or receiving thrombolysis or anticoagulant therapy;
8. Urine routine indicates urinary protein ≥ ++, or confirmed 24-hour urine protein ≥ 1.0 g;
9. Previously received radiotherapy, chemotherapy, hormonal therapy, surgery or molecular targeted therapy, after the completion of treatment (last dose), subjects less than 4 weeks before the study; adverse events caused by prior treatment (except for hair loss) did not recover To patients with ≤ CTCAE 1 degree;
10. There are significant clinically significant bleeding symptoms within 3 months before randomization or have a clear tendency to hemorrhage, such as gastrointestinal bleeding, active bleeding, baseline fecal occult blood + or above, or vasculitis;
11. Events of arteriovenous thrombosis occurring within 6 months prior to randomization, such as cerebrovascular accidents (including transient ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism;
12. Known hereditary or acquired bleeding and thrombophilia (eg hemophilia patients, coagulopathy, thrombocytopenia, hypersplenism, etc.);
13. The subject has an active infection;
14. Subjects with congenital or acquired immunodeficiency (such as HIV-infected patients), or active hepatitis (hepatitis B reference: HBsAg-positive and HBV DNA ≥ 104 copies/ml; hepatitis C reference: HCV antibody-positive);
15. Those who have used other drug clinical trials to study drugs within 4 weeks before the first dose;
16. The subject has had other malignant tumors within 5 years or at the same time (except for cured skin basal cell carcinoma and cervical carcinoma in situ and ovarian cancer);
17. Subjects have previously received other PD-1 antibody therapy or other immunotherapy against PD-1/PD-L1, or have previously received anti-angiogenic drugs (except Avastin);
18. Inoculate a live vaccine within less than 4 weeks of the study or possibly during the study period;
19. At the discretion of the investigator, the subject has other factors that may cause the study to be terminated midway. For example, other serious illnesses (including mental illness) require combined treatment, severe laboratory abnormalities, with family or Factors such as society can affect the safety of the subject.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rates (ORR) | up to two year
  the ratio of patients who are evaluated as CR or PR

SECONDARY OUTCOMES:
Duration of remission (DOR) | up to two year
  Defined as the time between the first assessment of a tumor as PR or CR and the first assessment as PD or any cause of death
Disease Control Rate (DCR) | up to two year
  It is defined as the proportion of patients whose tumors shrink or remain stable for a certain period of time, including CR, PR and SD.

CONTACTS AND LOCATIONS:
Overall Officials: Rui-Hua Xu, PhD, Study Chair — Sun Yat-sen University Cancer Hospital
Locations (1):
- Cancer center of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McDermott DF, Sosman JA, Sznol M, Massard C, Gordon MS, Hamid O, Powderly JD, Infante JR, Fasso M, Wang YV, Zou W, Hegde PS, Fine GD, Powles T. Atezolizumab, an Anti-Programmed Death-Ligand 1 Antibody, in Metastatic Renal Cell Carcinoma: Long-Term Safety, Clinical Activity, and Immune Correlates From a Phase Ia Study. J Clin Oncol. 2016 Mar 10;34(8):833-42. doi: 10.1200/JCO.2015.63.7421. Epub 2016 Jan 11. PMID 26755520